CLINICAL TRIAL: NCT02729311
Title: Paired Integrative Exercise Program for People With Dementia and Caregivers
Acronym: Paired PLIÉ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPSASA-15-364656
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Dementia
Keywords: exercise; function; quality of life; caregiver
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Paired PLIÉ Program
  Interventions: Behavioral: Paired PLIÉ Program
- Group 2 (Other): Waitlist control
  Interventions: Behavioral: Paired PLIÉ Program; Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Paired PLIÉ Program — The Paired PLIÉ Program is a novel, multimodal, movement program that focuses on abilities that are well maintained in people with dementia, including training procedural ('muscle') memory for basic daily movements, in-the-moment mindful body awareness, and social engagement. Group classes are held with affected individuals, care partners and instructors together. A monthly home visit also is provided.
Behavioral: Waitlist control — After engaging in usual activities for 12 weeks, the Waitlist control group participates in the Paired PLIÉ program.
  Arms: Group 2

SUMMARY:
Preventing Loss of Independence through Exercise (PLIÉ) is a unique, multimodal movement program for people with dementia (affected individuals) that is taught by trained instructors and combines physical, mental and social activities. The Paired PLIÉ Program is an adapted version designed for pairs of affected individuals and care partners. The goal of this study is to perform a randomized, controlled trial (RCT) with a delayed start design to examine the effects of the Paired PLIÉ Program on function and quality of life in affected individuals and care partners.

DETAILED DESCRIPTION:
Study participants are 30 pairs of individuals with mild-to-moderate dementia and their primary care partners (N=60 total) who are randomly assigned to Group 1 (immediate start) or Group 2 (delayed start). Pairs randomized to Group 1 participate together in the Paired PLIÉ program 2 days/week for 12 weeks (24 classes total) while pairs randomized to Group 2 continue with their usual activities. Then Group 1 transitions into a maintenance phase, and Group 2 participates in the Paired PLIÉ program 2 days/week for 12 weeks. Outcome data are collected in all study participants at baseline, mid-point and end-point so that we can examine the initial impact of the program as well as whether effects are maintained in Group 1. Outcome measures include cognitive function, physical performance, quality of life and caregiver well-being.

ELIGIBILITY:
Inclusion Criteria: Person with Cognitive Impairment

* diagnosis of cognitive impairment or dementia
* mild to moderate severity, defined as Clinical Dementia Rating of 0.5, 1 or 2
* willing and able to engage in study procedures
* English language fluency

Inclusion Criteria: Care Partner

* provide care for person with cognitive impairment
* willing and able to engage in study procedures
* English language fluency

Exclusion Criteria: Person with cognitive impairment

* planning to miss more than 2 weeks during the study period
* behavioral or physical issues that would be disruptive or dangerous to themselves or others (e.g., drug abuse, severe mental health issues)
* unable to take 2 steps independently without cane or walker
* terminal illness (life expectancy < 1 year)
* currently participating in another research study that could impact current study
* changes to dementia medications 3 months prior to baseline or changes planned during the study period

Exclusion Criteria: Care Partner

* planning to miss more than 2 weeks during the study period
* behavioral or physical issues that would be disruptive or dangerous to themselves or others (e.g., drug abuse, severe mental health issues)
* unable to take 2 steps independently without cane or walker
* terminal illness (life expectancy < 1 year)
* currently participating in another research study that could impact current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Barnes, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576
- [Background] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459
- [Background] Casey JJ, Harrison KL, Ventura MI, Mehling W, Barnes DE. An integrative group movement program for people with dementia and care partners together (Paired PLIE): initial process evaluation. Aging Ment Health. 2020 Jun;24(6):971-977. doi: 10.1080/13607863.2018.1553142. Epub 2019 Feb 12. PMID 30744387
- [Result] Mehling WE, Scott TM, Duffy J, Whitmer RA, Chesney MA, Boscardin WJ, Barnes DE. Dyadic Group Exercises for Persons with Memory Deficits and Care Partners: Mixed-Method Findings from the Paired Preventing Loss of Independence through Exercise (PLIE) Randomized Trial. J Alzheimers Dis. 2020;78(4):1689-1706. doi: 10.3233/JAD-200713. PMID 33185602
- See also: Facebook page — https://www.facebook.com/plie4dementia/
- See also: study website — http://plie4dementia.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited using a variety of strategies. We gave presentations at local caregiver support groups; distributed study flyers and brochures to psychiatrists, neurologists, and caregiver support managers; gave presentations at Medical Center Grand Rounds for attending physicians; and posted fliers in community settings and on social media (eg, Facebook).
Pre-assignment Details: Exclusion criteria were behavioral or physical issues that would be disruptive or dangerous to themselves or others (e.g., active psychosis, drug abuse, severe behavioral issues determined by interview); planning to move to a facility before the end of the study period; terminal illness (life expectancy.
Groups:
- Group 1: Paired PLIÉ Program, immediate start
  Paired PLIÉ Program: The Paired PLIÉ Program is a novel, multimodal, movement program that focuses on abilities that are well maintained in people with dementia, including training procedural ('muscle') memory for basic daily movements, in-the-moment mindful body awareness, and social engagement. Group classes are held with affected individuals, care partners and instructors together. A monthly home visit also is provided.
- Group 2: Waitlist control
  After engaging in usual activities for 12 weeks, the Waitlist control group participated in the Paired PLIÉ Program.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started (Participants were enrolled as dyads of persons with cognitive impairment (PWCI) + care partners (CPs).) | 30 | 30
Completed 12-week Assessment | 24 | 28
Completed | 22 | 28
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Population: 15 persons with cognitive impairment and 15 care partners per group
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This is for participants with cognitive impairment
  years
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 82.6 (6.0) | 77.3 (5.0) | 79.95 (5.5)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Care partners only
  years
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 71.6 (9.7) | 59.1 (17.4) | 60 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for persons with cognitive impairment and care partners analyzed separately
  Participants
    Participants with cognitive impairment: number analyzed (Participants) | 15 | 15 | 30
    Participants with cognitive impairment: Female | 7 | 9 | 16
    Participants with cognitive impairment: Male | 8 | 6 | 14
    Care partners: number analyzed (Participants) | 15 | 15 | 30
    Care partners: Female | 10 | 11 | 21
    Care partners: Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for persons with cognitive impairment and care partners analyzed separately
  Participants
    Persons with cognitive impairment: number analyzed (Participants) | 15 | 15 | 30
    Persons with cognitive impairment: American Indian or Alaska Native | 0 | 0 | 0
    Persons with cognitive impairment: Asian | 0 | 3 | 3
    Persons with cognitive impairment: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Persons with cognitive impairment: Black or African American | 1 | 3 | 4
    Persons with cognitive impairment: White | 14 | 8 | 22
    Persons with cognitive impairment: More than one race | 0 | 0 | 0
    Persons with cognitive impairment: Unknown or Not Reported | 0 | 1 | 1
    Care partners: number analyzed (Participants) | 15 | 15 | 30
    Care partners: American Indian or Alaska Native | 0 | 0 | 0
    Care partners: Asian | 0 | 3 | 3
    Care partners: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Care partners: Black or African American | 2 | 3 | 5
    Care partners: White | 12 | 8 | 20
    Care partners: More than one race | 0 | 0 | 0
    Care partners: Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30
Physical function (SPPB Score) PWCI - direct assessment [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery (SPPB) is a validated tool that provides an objective measure of physical performance in older adults. Tasks include tandem balance, usual walking speed, and chair stands. Scores may range from 0 to 12, with higher scores indicating better physical performance. Population: Measure administered only to persons with cognitive impairment. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 6.86 (2.66) | 6.53 (2.07) | 6.70 (2.37)
Quality of Life (QOL-AD) PWCI - self-report [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life in Alzheimer's Disease (QOL-AD) scale asks persons with cognitive impairment to rate their current quality of life on a 4-point Likert scale (poor, fair, good, excellent) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Internal consistency is excellent with a Cronbach's alpha coefficient of 0.82. Higher scores (range 4-52) indicate higher quality of life. Population: Data collected only in PWCI. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 40.21 (5.48) | 39.40 (5.33) | 39.81 (5.41)
Cognitive function (ADAS-cog) PWCI - direct assessment [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) was used to directly assess cognitive function in PWCI. It is one of the most commonly used outcome measures in dementia drug treatment trials. It includes direct assessment of learning (10-word list), naming (objects), following commands, constructional praxis (figure copying), ideational praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions. It has shown high consistency and test-retest reliability. Higher scores (range 0-70) indicate worse cognitive function. Population: Measure administered only to PWCI. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 32.21 (11.62) | 29.40 (9.38) | 30.81 (10.50)
Caregiver burden (CBI) CP - self-report [Mean (Standard Deviation); unit: units on a scale] — The Caregiver Burden Inventory (CBI) is a standard 24-item measure that includes questions about the CPs feelings about caregiving on a 5-point Likert scale with 5 domains. This measure has good internal consistency. Higher scores (range 0-96) indicate higher burden Population: Measure administered only to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 20.86 (9.04) | 26.93 (14.44) | 23.90 (11.74)
Balance score (SPPB) PWCI - direct assessment [Mean (Standard Deviation); unit: units on a scale] — Balance was assessed as part of the SPPB based on ability to stand with feet side-by-side together, in semi-tandem or tandem stance (range: ordinal variable 0-4). Higher scores indicate better performance Population: Measure only administered to PWCI. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 3.00 (1.30) | 2.80 (1.08) | 2.90 (1.19)
Independence (DAD) PWCI - CP report [Mean (Standard Deviation); unit: units on a scale] — The Disability Assessment for Dementia (DAD) is a standard measure that asks CPs to rate the participant's disability with 17 basic and 23 instrumental activities of daily living over the past 2 weeks. The DAD has high established validity and high test-retest reliability, inter-rater reliability, and internal consistency. Scores represent the percentage of activities performed independently during the past two weeks of those applicable (total number of questions answered yes/total questions applicable)∗100 with the range from 0 to 100. Higher scores indicate greater independence. Population: Measure only administered to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 69.98 (22.96) | 64.60 (29.28) | 67.29 (26.12)
Falls Efficacy (FES) PWCI - self-report [Mean (Standard Deviation); unit: units on a scale] — Participants were asked about their concern about falling doing 10 activities. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy). Population: Data analyzed separately for PWCI and CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 12.43 (3.44) | 12.87 (5.55) | 12.65 (4.5)
Falls Efficacy (FES) PWCI - CP report [Mean (Standard Deviation); unit: units on a scale] — Care partners were asked about their concern that participants with cognitive impairment might fall doing 10 activities. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy). Population: Data analyzed separately for PWCI and CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 14.07 (5.09) | 16.00 (6.49) | 15.04 (5.79)
Caregiving (PAC) CP - self-report [Mean (Standard Deviation); unit: units on a scale] — The Positive Aspects of Caregiving (PAC) scale includes 9 questions about the benefits of caregiving noticed by the CPs about themselves, which are rated on a 5-point Likert scale. This measure has high internal consistency and can improve with CP training interventions.
  Total scores range from 11 to 55 with higher scores indicating more positive feelings. Population: Measure only administered to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 41.93 (5.97) | 43.67 (9.10) | 42.8 (7.54)
Quality of life (QOL-AD) PWCI - CP report [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Scale in Alzheimer's Disease (QOL-AD) also asks CPs to rate the current quality of life for PWCI on a 4-point Likert scale. Higher scores (range 4-52) indicate higher quality of life. Population: Data analyzed separately for PWCI and CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 35.86 (3.37) | 34.40 (4.64) | 35.13 (4.01)
Behaviors - frequency (NPI-N) PWCI - CP report [Mean (Standard Deviation); unit: units on a scale] — Neuropsychiatric Inventory - Number (NPI-N) asks CPs about the presence of dementia-related behaviors in PWCI. Scores may range from 0-12. Higher scores indicate more behaviors. Population: Measure only administered to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 2.64 (1.95) | 4.20 (3.12) | 3.42 (2.54)
Behaviors - severity (NPI-FS) PWCI - CP report [Mean (Standard Deviation); unit: units on a scale] — Neuropsychiatric Inventory - Frequency/Severity (NPI-FS) asks CPs to rate the frequency and severity of dementia-related behaviors. Scores may range from 0-144 and are calculated by multiplying frequency by severity of behaviors. Higher scores indicate greater frequency/severity. Population: Measure only administered to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 7.57 (6.17) | 13.57 (14.90) | 10.57 (10.54)
Behaviors - distress (NPI-CD) CP - self-report [Mean (Standard Deviation); unit: units on a scale] — Neuropsychiatric Inventory - Caregiver Distress (NPI-CD) asks CPs to rate their feelings of distress associated with dementia-related behaviors. Scores may range from 0-60. Higher scores indicate greater distress. Population: Measure only administered to CPs. Data missing for 1 person who withdrew before baseline.
  units on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 4.29 (3.43) | 9.73 (12.29) | 7.01 (7.86)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function (PWCI, Direct Assessment)
Description: Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) - total score This was was used to directly assess cognitive function in PWCI. It is one of the most commonly used outcome measures in dementia drug treatment trials. It includes direct assessment of learning (10-word list), naming (objects), following commands, constructional praxis (figure copying), ideational praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions. The ADAS-cog has shown high consistency and test-retest reliability. Higher scores (range 0-70) indicate worse cognitive function.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 2: Paired PLIÉ Program, delayed start
  Paired PLIÉ Program: The Paired PLIÉ Program is a novel, multimodal, movement program that focuses on abilities that are well maintained in people with dementia, including training procedural ('muscle') memory for basic daily movements, in-the-moment mindful body awareness, and social engagement. Group classes are held with affected individuals, care partners and instructors together. A monthly home visit also is provided.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 31.78 (11.15) | 32.60 (13.62)

2. Primary Outcome: Physical Function (Affected Individual, Direct Assessment)
Description: Short Physical Performance Battery (SPPB) - total score The Short Physical Performance Battery (SPPB) was developed by the National Institute on Aging to provide an objective tool for measuring physical performance in older adults. It includes direct assessment of lower body strength, balance and gait speed that provide a summary score (range 0-12). Higher scores indicate higher performance ability.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 6.50 (2.32) | 6.57 (2.50)

3. Primary Outcome: Quality of Life (Affected Individual, Self-report)
Description: Quality of life in Alzheimer's disease (QOL-AD) - total score The Quality of Life Scale in Alzheimer's Disease (QOL-AD) asks PWDs to rate their current quality of life on a 4-point Likert scale (poor, fair, good, excellent) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Internal consistency is excellent with a Cronbach's alpha coefficient of 0.82. Higher scores (range 4-52) indicate higher quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 41.42 (4.74) | 40.14 (5.80)

4. Primary Outcome: Caregiver Burden (Caregiver, Self-report)
Description: Caregiver Burden Inventory (CBI) - total score This is a standard 24-item measure that includes questions about the CPs feelings about caregiving on a 5-point Likert scale with 5 domains. This measure has good internal consistency. Higher scores (range 0-96) indicate higher burden.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 23.27 (11.20) | 28.85 (16.67)

5. Primary Outcome: Cognitive Function (Affected Individual, Direct Assessment)
Description: Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) - total score The Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) was used to directly assess cognitive function in PWD. It is one of the most commonly used outcome measures in dementia drug treatment trials. It includes direct assessment of learning (10-word list), naming (objects), following commands, constructional praxis (figure copying), ideational praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions. The ADAS-cog has shown high consistency and test-retest reliability. Higher scores (range 0-70) indicate worse cognitive function.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 30.97 (11.46) | 32.67 (11.48)

6. Primary Outcome: Physical Function (Affected Individual, Direct Assessment)
Description: as for outcome 2
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 6.70 (2.26) | 6.69 (2.36)

7. Primary Outcome: Quality of Life (Affected Individual, Self-report)
Description: Quality of life in Alzheimer's disease (QOL-AD) - total score Quality of life in Alzheimer's disease (QOL-AD) - total score The Quality of Life Scale in Alzheimer's Disease (QOL-AD) asks PWDs to rate their current quality of life on a 4-point Likert scale (poor, fair, good, excellent) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Internal consistency is excellent with a Cronbach's alpha coefficient of 0.82. Higher scores (range 4-52) indicate higher quality of life.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 41.20 (5.45) | 40.85 (5.81)

8. Primary Outcome: Caregiver Burden (Caregiver, Self-report)
Description: Caregiver Burden Inventory (CBI) - total score Caregiver Burden Inventory (CBI) - total score This is a standard 24-item measure that includes questions about the CPs feelings about caregiving on a 5-point Likert scale with 5 domains. This measure has good internal consistency. Higher scores (range 0-96) indicate higher burden.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 27.33 (12.73) | 30.00 (16.64)

9. Secondary Outcome: Independence (Affected Individual, Caregiver Report)
Description: Disability Assessment for Dementia (DAD) - total score Independence (PWD - CP report). The Disability Assessment for Dementia (DAD)is a standard measure that asks CPs to rate the participant's disability with 17 basic and 23 instrumental activities of daily living over the past 2 weeks. The DAD has high established validity and high test-retest reliability, inter-rater reliability, and internal consistency. Scores represent the percentage of activities performed independently during the past two weeks of those applicable (total number of questions answered yes/total questions applicable)∗100 with the range from 0 to 100. Higher scores indicate greater independence
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 23.27 (11.20) | 28.85 (16.67)

10. Secondary Outcome: Dementia-related Behaviors - Number (Affected Individual, Caregiver Report)
Description: The Neuropsychiatric Inventory (NPI) was administered to assess the number (NPI-N), caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, and appetite/eating) by CP report and has good test-retest reliability and internal consistency. NPI-N scores range from 0-12. Higher scores indicate worse outcomes (i.e., more behaviors, greater frequency/severity and greater distress).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 2.25 (1.82) | 4.43 (3.06)

11. Secondary Outcome: Dementia-related Behaviors - Severity (Affected Individual, Caregiver Report)
Description: Neuropsychiatric Inventory (NPI) - total frequency * severity measures distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, and appetite/eating) by CP report and has good test-retest reliability and internal consistency. NPI-FS was calculated by multiplying the frequency∗severity of behaviors, which had a range of 0-144. Higher scores indicate worse outcomes (i.e., more behaviors, greater frequency/severity and greater distress).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 6.50 (7.60) | 15.69 (16.03)

12. Secondary Outcome: Dementia-related Behaviors - Caregiver Distress (Caregiver, Self-report)
Description: Neuropsychiatric Inventory (NPI) - total distress level of caregiver distress (NPI-CD) caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, and appetite/eating) by CP report and has good test-retest reliability and internal consistency. NPI-CD range from 0-60. Higher scores indicate worse outcomes (i.e., more behaviors, greater frequency/severity and greater distress).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 4.58 (5.00) | 11.21 (12.58)

13. Secondary Outcome: Falls Efficacy (Affected Individual, Self-report)
Description: Falls Efficacy Scale (FES) - total score We administered a modified version of the Falls Efficacy Scale (FES) to assess concern about falling for the PWD in 10 different scenarios. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy). Although the FES has been validated in individuals with cognitive impairment the questionnaire was administered separately to PWD and CPs to obtain their independent perspetive
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 13.58 (5.35) | 12.86 (5.33)

14. Secondary Outcome: Falls Efficacy (Affected Individual, Caregiver Report)
Description: Falls Efficacy Scale (FES) - total score We administered a modified version of the Falls Efficacy Scale (FES) to assess concern about falling for the PWD in 10 different scenarios. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy). Although the FES has been validated in individuals with cognitive impairment the questionnaire was administered separately to PWD and CPs to obtain their independent perspective
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 14.17 (5.87) | 15.29 (7.76)

15. Secondary Outcome: Quality of Life (Affected Individual, Caregiver Report)
Description: Quality of Life in Alzheimer's Disease (QOL-AD) - total score The Quality of Life Scale in Alzheimer's Disease (QOL-AD) also asks CPs to rate the PWD current quality of life on the same scale as the PWD QOL self-report. It asks to rate their current quality of life on a 4-point Likert scale (poor, fair, good, excellent) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Internal consistency is excellent with a Cronbach's alpha coefficient of 0.82. Higher scores (range 4-52) indicate higher quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 35.42 (4.29) | 33.00 (7.12)

16. Secondary Outcome: Mood (Caregiver, Self-report)
Description: Geriatric Depression Scale (GDS) - total score. The Geriatric Depression Scale (GDS) is a standard measure that includes 15 yes/no questions assessing depressive symptomatology over the past week. PWD and CP answered separately regarding their own mood. This scale ranges from 0 to 15 and has been validated in people with and without cognitive impairment. Higher scores indicate more depressive symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 1.92 (1.88) | 2.69 (2.14)

17. Secondary Outcome: Feelings About Caregiving (Caregiver, Self-report)
Description: Positive Aspects of Caregiving (PAC) - total score. The PAC scale includes 9 questions about the benefits of caregiving noticed by the CPs about themselves, which are rated on a 5-point Likert scale. This measure has high internal consistency and can improve with CP training interventions. Total scores range from 11 to 55 with higher scores indicating more positive feelings.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
units on a scale | 43.50 (7.20) | 44.07 (7.68)

18. Secondary Outcome: Independence (Affected Individual, Caregiver Report)
Description: Disability Assessment for Dementia (DAD) - total score. The DAD is a standard measure that asks CPs to rate the participant's disability with 17 basic and 23 instrumental activities of daily living over the past 2 weeks. The DAD has high established validity and high test-retest reliability, inter-rater reliability, and internal consistency. Scores represent the percentage of activities performed independently during the past two weeks of those applicable (total number of questions answered yes/total questions applicable)∗100 with the range from 0 to 100. Higher scores indicate greater independence.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of independence activities
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
percentage of independence activities | 64.05 (24.97) | 59.04 (32.15)

19. Secondary Outcome: Dementia-related Behaviors - Number (Affected Individual, Caregiver Report)
Description: Neuropsychiatric Inventory (NPI) - total number of symptoms. The NPI asks CPs to report the number (NPI-N), frequency/severity (NPI-FS), and level of caregiver distress (NPI-CD) caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, and appetite/eating) and has good test-retest reliability and internal consistency. NPI-N scores range from 0-12.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: count of symptoms
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
count of symptoms | 2.20 (2.15) | 3.93 (3.12)

20. Secondary Outcome: Dementia-related Behaviors - Frequency and Severity (Affected Individual, Caregiver Report)
Description: Neuropsychiatric Inventory - Frequency/Severity (NPI-FS). For each behavior present, care partners are asked to rate the frequency (occasionally=1, often=2, frequently=3, very frequently=4) and severity (mild=1, moderate=2, severe=3). The score is obtained by multiplying frequency and severity and adding them for each behavior. Scores may range from 0 to 144 with higher scores indicating more frequent/severe behaviors.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 4.67 (5.48) | 12.54 (11.16)

21. Secondary Outcome: Dementia-related Behaviors - Caregiver Distress (Caregiver, Self-report)
Description: Neuropsychiatric Inventory - caregiver distress (NPI-CD). For each behavior, caregivers are asked how emotionally distressing they find the behavior on a scale from 0 (not distressing at all) to 5 (extreme or very severe). Scores may range from 0 to 60 with higher scores indicating greater distress.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 4.70 (6.58) | 9.64 (10.68)

22. Secondary Outcome: Falls Efficacy (Affected Individual, Self-report)
Description: Falls Efficacy Scale (FES) - total score. We administered a modified version of the FES to assess the participant's concern about falling in 10 different scenarios. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 13.40 (4.48) | 15.93 (9.22)

23. Secondary Outcome: Falls Efficacy (Affected Individual, Caregiver Report)
Description: Falls Efficacy Scale (FES) - total score. We administered a modified version of the FES to assess the caregiver's concern about the participant falling in 10 different scenarios. Response categories used a 4-point Likert scale (range: 10 to 40), with higher scores indicating greater concern about falling (i.e., lower efficacy).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 16.00 (7.13) | 16.14 (6.70)

24. Secondary Outcome: Quality of Life (Person With Dementia, Caregiver Report)
Description: Quality of Life in Alzheimer's Disease (QOL-AD) - total score. Caregivers were asked to rate the QOL of participants with dementia on a 4-point Likert scale (poor, fair, good, excellent) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Internal consistency is excellent with a Cronbach's alpha coefficient of 0.82. Higher scores (range 4-52) indicate higher quality of life.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 32.50 (4.58) | 32.93 (7.31)

25. Secondary Outcome: Mood (Caregiver, Self-report)
Description: Geriatric Depression Scale (GDS) - total score. The GDS is a standard measure that includes 15 yes/no questions assessing depressive symptomatology over the past week. PWD and CP answered separately regarding their own mood. This scale ranges from 0 to 15 and has been validated in people with and without cognitive impairment. Higher scores indicate more depressive symptoms.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 2.22 (1.20) | 2.57 (2.77)

26. Secondary Outcome: Feelings About Caregiving (Caregiver, Self-report)
Description: Positive Aspects of Caregiving (PAC) - total score. The PAC includes 9 questions about the benefits of caregiving noticed by the CPs about themselves, which are rated on a 5-point Likert scale. This measure has high internal consistency and can improve with CP training interventions. Total scores range from 11 to 55 with higher scores indicating more positive feelings.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 15
score on a scale | 39.33 (6.04) | 42.93 (8.41)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: We asked caregivers to report any major health-related events or falls in themselves or the person with cognitive impairment through monthly telephone check-in calls.
Groups:
- Group 1 - Persons With Cognitive Impairment: Paired PLIÉ Program, immediate start - persons with cognitive impairment
- Group 1 - Caregivers: Paired PLIÉ Program, immediate start - caregivers
- Group 2 - Persons With Cognitive Impairment: Waitlist control, delayed start - persons with cognitive impairment
- Group 2 - Caregivers: Waitlist control, delayed start - caregivers
Arm/Group | Group 1 - Persons With Cognitive Impairment | Group 1 - Caregivers | Group 2 - Persons With Cognitive Impairment | Group 2 - Caregivers
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15 | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/15 | 4/15 | 5/15 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Persons With Cognitive Impairment (N=15) | Group 1 - Caregivers (N=15) | Group 2 - Persons With Cognitive Impairment (N=15) | Group 2 - Caregivers (N=15)
Emergency visit or hospitalization (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Persons With Cognitive Impairment (N=15) | Group 1 - Caregivers (N=15) | Group 2 - Persons With Cognitive Impairment (N=15) | Group 2 - Caregivers (N=15)
Falls / Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 4 (4) | 1 (1)
Other AEs (General disorders) | 2 (2) | 4 (4) | 1 (2) | 0 (0) — Includes infections, gastrointestinal issues, and psychiatric issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT02729311/Prot_SAP_000.pdf